CLINICAL TRIAL: NCT07026409
Title: Study of Epilepsy and Seizure in Elderly Patients in Sohag University Hospitals.
Brief Title: This Study Will Assess the Etiology, Potential Risk Factors, and Seizure Types in Patients Over 50 With Epileptic Seizure Disorder, Using Laboratory Tests, EEG, and Neuroimaging Findings.
Status: Active, not recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mostafa Elsayed Abdelwahab, Resident at Department of Neurology and Psychological Medicine Sohag university hospital., Sohag University
Other Study IDs: Soh-Med--25-5-3MS
Record Dates: First submitted 2025-06-03; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-05

CONDITIONS: Epilepsy
Keywords: Epilepsy,Elderly,Seizure,EEG.
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study underscores the importance of studying the etiology, clinical characteristics, and types of epilepsy in the elderly to improve diagnosis and management in our community.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of epilepsy and epileptic seizures will be clinically established based on patient history, following the Glossary of Descriptive Terminology for Ictal Semiology by the International League Against Epilepsy (ILAE) Task Force on Classification and Terminology, as well as the Operational Classification of Seizure Types (ILAE, 2017).

Exclusion Criteria:

* • Inability to determine the onset of epilepsy or epileptic seizures, or a history of seizures occurring before the age of 50.

  * Metabolic disturbances such as hypoglycemia, uremia, or electrolyte imbalances.
  * Patients who refuse to participate in the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include all consecutive patients aged 50 years and older who are admitted to the inpatient Neuropsychiatry Department or attend the Epilepsy Specialized Outpatient Clinic at Sohag University Hospital with epilepsy or new-onset epileptic .
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Risk factors of epilepsy in elderly | Baseline
  MRI brain for structural or pathological abnormalities
Etiology of epilepsy in elderly | Baseline
  Electroencephalography for electrical changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Sohag University, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided